CLINICAL TRIAL: NCT03151395
Title: Occurrence of Potential Bacterial and Viral Pathogens in Stable Chronic Obstructive Pulmonary Disease (COPD) and During Acute Exacerbations of COPD (AECOPD), in Asia Pacific
Brief Title: Occurrence of Potential Bacterial and Viral Pathogens in Stable Chronic Obstructive Pulmonary Disease and During Acute Exacerbations of the Disease, in Asia Pacific
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201112
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Disorders
Keywords: COPD; AECOPD; GOLD (Global Initiative for Chronic Obstructive Lung Disease); Asia Pacific
MeSH Terms: conditions — Respiration Disorders; Pulmonary Disease, Chronic Obstructive | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total Group (Other): Moderate to very severe Chronic Obstructive Pulmonary Disease (COPD) patients with at least 1 documented moderate or severe Acute exacerbation of COPD (AECOPD) in the year before enrolment and for whom sputum and blood samples are collected during specified visits
  Interventions: Other: Sputum and blood sampling

INTERVENTIONS:
Other: Sputum and blood sampling — Evaluation of the occurrence of potential bacterial and viral pathogens in the sputum of stable COPD patients and at the time of AECOPD.

SUMMARY:
Since the infectious aetiology of AECOPD has been suggested to vary according to geographical region, the primary purpose of this study (which will be conducted in several countries in Asia Pacific) is to evaluate the occurrence of bacterial and viral pathogens in the sputum of stable COPD patients and at the time of AECOPD. Given the increasing and projected burden of COPD in the Asia Pacific region, this study will also evaluate the frequency, severity and duration of AECOPD, as well as the impact of AECOPD on health-related quality of life (HRQOL), healthcare utilisation and lung function.

DETAILED DESCRIPTION:
The protocol has been amended to implement the following changes:

* Alignment of the protocol to the updated GOLD consensus report of 2017 and the COPD fact sheet.
* Alignment of the study endpoints to the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of electronic Diary Card, sputum sampling, pre- and post-bronchodilator spirometry, return for follow-up visits).
* Written informed consent obtained from the subject.
* Male or female aged 40 years or older at the time of enrolment.
* Confirmed diagnosis of moderate to very severe COPD based on post-bronchodilator spirometry (i.e. forced expiratory volume in 1 second [FEV1] over forced vital capacity [FVC] ratio [FEV1/ FVC] < 0.7 and FEV1 < 80% predicted [GOLD grades 2, 3 and 4].
* Stable COPD patient* with documented history** (e.g. medical record verification) of at least 1 moderate or severe AECOPD within the 12 months before study entry.

  * Patient for whom the last episode of AECOPD is resolved for at least 30 days at the time of study entry.

    * Note: A documented history of a COPD exacerbation (e.g., medical record verification) is a medical record of worsening COPD symptoms that required systemic/oral corticosteroids and/or antibiotics (for a moderate exacerbation) or hospitalization (for a severe exacerbation). Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnea, sputum volume, or sputum purulence (color). Subject verbal reports are not acceptable.
* Current or former tobacco smoker (cigarette) with a smoking history of ≥ 10 pack-years OR a subject exposed to biomass smoke for ≥ 20 years.
* Able to provide a sputum sample at Screening Visit.

Exclusion Criteria:

* Diagnosed with a respiratory disorder other than COPD (such as sarcoidosis, active tuberculosis or receiving tuberculosis treatment, clinically significant bronchiectasis, lung fibrosis, pulmonary embolism, pneumothorax, lung cancer diagnosed within the previous 5 years, current primary diagnosis of asthma in the opinion of the investigator), or chest X-ray revealing evidence of clinically significant abnormalities not believed to be due to the presence of COPD*. Subjects with allergic rhinitis do not need to be excluded and may be enrolled at the discretion of the investigator.

  * A chest X-ray must be taken at Screening Visit, if no chest X-ray taken within the previous 3 months is available.
* Diagnosis of α-1 antitrypsin deficiency as the underlying cause of COPD.
* Undergone or has had lung surgery 12 months before, or plans to have lung surgery 12 months after, study entry.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Received chemotherapy within the 12 months before study entry.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/ product (pharmaceutical product or device).
* Administration of antibiotics within 1 month of study entry OR continuous administration of antibiotics (defined as more than 30 days in total) within 90 days before study entry.
* Systemic administration of corticosteroids for more than 14 consecutive days within 90 days prior to informed consent.
* Contraindication for spirometry testing (such as recent eye surgery, recent thoracic or abdominal surgery procedures, unstable cardiovascular status, recent myocardial infarction or pulmonary embolism).
* Psychiatric illness or any other condition that interferes with the ability to understand the study procedures.
* Pregnant female.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Hong Kong (3):
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Lai Chi Kok
  - GSK Investigational Site, Shatin
- Philippines (4):
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Jaro, Iloilo City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Marilao, Bulacan
- South Korea (4):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Gangwon-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Taiwan (4):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Keelung
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei

REFERENCES:
- [Derived] Taddei L, Malvisi L, Hui DS, Malvaux L, Samoro RZ, Lee SH, Yeung YC, Liu YC, Arora AK. Airway pathogens detected in stable and exacerbated COPD in patients in Asia-Pacific. ERJ Open Res. 2022 Sep 26;8(3):00057-2022. doi: 10.1183/23120541.00057-2022. eCollection 2022 Jul. PMID 36171985

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Group
Started | 197
Completed | 182
Not Completed | 15
Not completed — Adverse Event | 2
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 6
Not completed — Subjects could not perform last visit before study completion date due to local COVID19 restrictions | 3
Not completed — Unspecified reason | 4

BASELINE CHARACTERISTICS:
Arm/Group | Total Group
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 187
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - EAST ASIAN HERITAGE | 126
  ASIAN - SOUTH EAST ASIAN HERITAGE | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Sputum Samples Positive for Bacterial Pathogens as Identified by Bacteriological Methods, in Any Stable COPD Patients and During AECOPDs
Description: The proportion of sputum samples obtained at each visit (confirmed stable or AECOPD visits) and positive for specific bacterial pathogens by bacteriological methods (overall and by bacterial species). Numerator is the number of sputum samples positive for a given pathogen and denominator is the number of visits with a sputum sample tested for a given pathogen. Proportion is computed with 95% confidence intervals. A confirmed stable visit is defined as a scheduled study visit for which the investigator confirms that the subject is stable/ has recovered from a previous exacerbation. Bacterial pathogens include Haemophilus influenzae (Hi), Non-typeable Haemophilus influenzae (NTHi), non-Haemophilus influenzae (Non-Hi), Moraxella catarrhalis (M. catarrhalis), Streptococcus pneumoniae (S. pneumoniae), Staphylococcus aureus (S. aureus), Pseudomonas aeruginosa (P. aeruginosa), Klebsiella pneumoniae (K. pseumoniae), Acinetobacter baumannii (A. baumannii).
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: Analysis was performed on the Full Analysis Set which included all screened subjects who were enrolled except for those subjects who discontinued the study at Month 0 visit.
Measure: Number (95% Confidence Interval); unit: Percentage of sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 196
Percentage of sputum samples
  Any, Any stable visit | 74.2 [70.4 to 77.7]
  Any, Any AECOPD visit: number analyzed (Participants) | 88
  Any, Any AECOPD visit | 78 [72.1 to 83.2]
  Hi, Any stable visit: number analyzed (Participants) | 29
  Hi, Any stable visit | 94.6 [84.2 to 99.1]
  Hi, Any AECOPD visit: number analyzed (Participants) | 13
  Hi, Any AECOPD visit | 94.1 [76.6 to 99.7]
  NTHi, Any stable visit: number analyzed (Participants) | 29
  NTHi, Any stable visit | 94.6 [84.2 to 99.1]
  NTHi, Any AECOPD visit: number analyzed (Participants) | 13
  NTHi, Any AECOPD visit | 94.1 [76.6 to 99.7]
  Non-Hi, Any stable visit: number analyzed (Participants) | 29
  Non-Hi, Any stable visit | 5.4 [0.9 to 15.8]
  Non-Hi, Any AECOPD visit: number analyzed (Participants) | 13
  Non-Hi, Any AECOPD visit | 5.9 [0.3 to 23.4]
  M. catarrhalis, Any stable visit | 0.9 [0.3 to 1.9]
  M. catarrhalis, Any AECOPD visit: number analyzed (Participants) | 88
  M. catarrhalis, Any AECOPD visit | 3.3 [1.5 to 6.4]
  S. pneumoniae, Any stable visit | 2.5 [1.4 to 4.1]
  S. pneumoniae, Any AECOPD visit: number analyzed (Participants) | 88
  S. pneumoniae, Any AECOPD visit | 2.4 [0.9 to 5.1]
  S. aureus, Any stable visit | 3.1 [1.8 to 4.7]
  S. aureus, Any AECOPD visit: number analyzed (Participants) | 88
  S. aureus, Any AECOPD visit | 3.3 [1.5 to 6.4]
  P. aeruginosa, Any stable visit | 8.5 [6.4 to 11.0]
  P. aeruginosa, Any AECOPD visit: number analyzed (Participants) | 88
  P. aeruginosa, Any AECOPD visit | 14.4 [10.0 to 19.5]
  K. pneumoniae, Any stable visit | 26.4 [22.8 to 30.1]
  K. pneumoniae, Any AECOPD visit: number analyzed (Participants) | 88
  K. pneumoniae, Any AECOPD visit | 24.9 [19.3 to 31.0]
  A. baumannii, Any stable visit | 2.2 [1.2 to 3.6]
  A. baumannii, Any AECOPD visit: number analyzed (Participants) | 88
  A. baumannii, Any AECOPD visit | 4.3 [2.1 to 7.6]
  Other bacteria, Any stable visit | 47.7 [43.5 to 51.8]
  Other bacteria, Any AECOPD visit: number analyzed (Participants) | 88
  Other bacteria, Any AECOPD visit | 45 [38.3 to 51.8]

2. Primary Outcome: Percentage of Sputum Samples Positive for Viral Pathogens as Identified by Polymerase Chain Reaction (PCR) in Stable COPD Patients and During AECOPDs
Description: The proportion of sputum samples obtained at each visit (confirmed stable visits and AECOPD visits) and positive for specific viral pathogens by PCR (overall and by viral species). The numerator is the number of sputum samples positive for a given pathogen and the denominator is the number of visits with a sputum sample tested for a given pathogen. The proportion is calculated with 95% confidence intervals. Viral pathogens, as identified by PCR, include respiratory syncytial virus (RSV), parainfluenza virus, enterovirus, human rhinovirus (HRV), metapneumovirus, influenza virus, adenovirus, bocavirus and coronavirus.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 195
Percentage of sputum samples
  Any, Any stable visit | 15 [12.2 to 18.2]
  Any, Any AECOPD visit: number analyzed (Participants) | 88
  Any, Any AECOPD visit | 35.6 [29.1 to 42.5]
  RSV, Any stable visit | 0.9 [0.3 to 2.0]
  RSV, Any AECOPD visit: number analyzed (Participants) | 88
  RSV, Any AECOPD visit | 1 [0.2 to 3.1]
  Parainfluenza virus, Any stable visit | 0.7 [0.2 to 1.7]
  Parainfluenza virus, Any AECOPD visit: number analyzed (Participants) | 88
  Parainfluenza virus, Any AECOPD visit | 4.7 [2.3 to 8.2]
  Enterovirus, Any stable visit | 0.6 [0.1 to 1.4]
  Enterovirus, Any AECOPD visit: number analyzed (Participants) | 88
  Enterovirus, Any AECOPD visit | 0 [0.0 to 1.9]
  HRV, Any stable visit | 8.1 [6.0 to 10.6]
  HRV, Any AECOPD visit: number analyzed (Participants) | 88
  HRV, Any AECOPD visit | 16.6 [11.8 to 22.3]
  Metapneumovirus, Any stable visit | 0 [0.0 to 0.7]
  Metapneumovirus, Any AECOPD visit: number analyzed (Participants) | 88
  Metapneumovirus, Any AECOPD visit | 0 [0.0 to 1.9]
  Influenza virus, Any stable visit | 0.7 [0.2 to 1.7]
  Influenza virus, Any AECOPD visit: number analyzed (Participants) | 88
  Influenza virus, Any AECOPD visit | 8.2 [4.9 to 12.7]
  Adenovirus, Any stable visit | 2 [1.1 to 3.4]
  Adenovirus, Any AECOPD visit: number analyzed (Participants) | 88
  Adenovirus, Any AECOPD visit | 4.1 [1.9 to 7.6]
  Bocavirus, Any stable visit | 0.2 [0.0 to 0.8]
  Bocavirus, Any AECOPD visit: number analyzed (Participants) | 88
  Bocavirus, Any AECOPD visit | 0 [0.0 to 1.9]
  Coronavirus, Any stable visit | 2.6 [1.5 to 4.1]
  Coronavirus, Any AECOPD visit: number analyzed (Participants) | 88
  Coronavirus, Any AECOPD visit | 5.7 [3.0 to 9.5]

3. Secondary Outcome: Percentage of Sputum Samples Positive for Bacterial Pathogens in Stable COPD Patients and During AECOPDs, as Identified by PCR
Description: The proportion of sputum samples obtained at each confirmed stable/AECOPD visit and positive for specific bacterial pathogens as measured by real-time qualitative PCR/quantitative PCR, (overall and by bacterial species,) are computed with 95% confidence intervals. The numerator is the number of sputum samples positive for a given pathogen and the denominator is the number of visits with a sputum sample tested for a given pathogen. The bacterial pathogens include H. influenzae, M. catarrhalis, S. pneumoniae, S. aureus, P. aeruginosa and S. pyogenes. A confirmed stable visit is defined as a scheduled study visit for which the investigator confirms that the subject is stable / has recovered from a previous exacerbation.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 195
Percentage of sputum samples
  Any, Any stable visit | 67 [63.0 to 70.9]
  Any, Any AECOPD visit: number analyzed (Participants) | 88
  Any, Any AECOPD visit | 74.7 [68.3 to 80.5]
  H. influenzae, Any stable visit | 42.9 [38.7 to 47.0]
  H. influenzae, Any AECOPD visit: number analyzed (Participants) | 88
  H. influenzae, Any AECOPD visit | 39.7 [33.0 to 46.7]
  M. catarrhalis, Any stable visit | 13.7 [11.0 to 16.8]
  M. catarrhalis, Any AECOPD visit: number analyzed (Participants) | 88
  M. catarrhalis, Any AECOPD visit | 26.8 [20.9 to 33.3]
  S. pneumoniae, Any stable visit | 16.8 [13.9 to 20.1]
  S. pneumoniae, Any AECOPD visit: number analyzed (Participants) | 88
  S. pneumoniae, Any AECOPD visit | 19.1 [14.0 to 25.0]
  S. aureus, Any stable visit | 10.6 [8.2 to 13.4]
  S. aureus, Any AECOPD visit: number analyzed (Participants) | 88
  S. aureus, Any AECOPD visit | 9.3 [5.7 to 13.9]
  P. aeruginosa, Any stable visit | 16.3 [13.4 to 19.6]
  P. aeruginosa, Any AECOPD visit: number analyzed (Participants) | 88
  P. aeruginosa, Any AECOPD visit | 16.5 [11.7 to 22.1]
  S. pyogenes, Any stable visit | 0.4 [0.1 to 1.1]
  S. pyogenes, Any AECOPD visit: number analyzed (Participants) | 88
  S. pyogenes, Any AECOPD visit | 1 [0.2 to 3.1]

4. Secondary Outcome: Number of Sputum Samples in a Given Category Relative to All Combinations for Each Bacterial Pathogen, When Identified by Bacteriological Methods or PCR, at Any Visit
Description: Concordance between bacteriological methods (culture) and PCR sputum results are described for all the combinations of bacterial presence by both measures. Each category name includes the following parameters: Bacteria species-Culture (yes/no)- PCR (yes/no). Concordance is expressed as the number of sputum samples in a given category among the total number of sputum samples assessed for the presence of bacterial pathogens by both culture and PCR
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: Analysis was performed on the sputum samples taken from Full Analysis Set which included all screened subjects who were enrolled except for those subjects who discontinued the study at Month 0 visit.
Measure: Count of Units; unit: Sputum samples
Units Other Than Participants: Sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 197
Number analyzed (Sputum samples) | 740
Sputum samples
  H. influenzae, Culture No, PCR No | 425
  H. influenzae, Culture No, PCR Yes | 260
  H. influenzae, Culture Yes, PCR No | 4
  H. influenzae, Culture Yes, PCR Yes | 51
  M. catarrhalis, Culture No, PCR No | 613
  M. catarrhalis, Culture No, PCR Yes | 115
  M. catarrhalis, Culture Yes, PCR No | 0
  M. catarrhalis, Culture Yes, PCR Yes | 12
  S. pneumoniae, Culture No, PCR No | 610
  S. pneumoniae, Culture No, PCR Yes | 111
  S. pneumoniae, Culture Yes, PCR No | 1
  S. pneumoniae, Culture Yes, PCR Yes | 18
  S. aureus, Culture No, PCR No | 655
  S. aureus, Culture No, PCR Yes | 62
  S. aureus, Culture Yes, PCR No | 9
  S. aureus, Culture Yes, PCR Yes | 14
  P. aeruginosa, Culture No, PCR No | 599
  P. aeruginosa, Culture No, PCR Yes | 67
  P. aeruginosa, Culture Yes, PCR No | 20
  P. aeruginosa, Culture Yes, PCR Yes | 54

5. Secondary Outcome: Number of Sputum Samples Positive for Bacterial Pathogens (Overall and by Species) in Stable COPD Patients, as Identified by Bacteriological Methods, and Classified by Global Initiative for Chronic Obstructive Lung Disease (GOLD) Grade
Description: Number of sputum samples obtained at each confirmed stable visit, and positive for bacterial pathogens by bacteriological methods (overall and by bacterial species). The spirometric classification of airflow limitation in COPD patients is based on post-bronchodilator forced expiratory volume in 1 second (FEV1) and can be divided into four GOLD grades [GOLD, 2013]: GOLD 1 (MILD): FEV1 ≥ 80% predicted; GOLD 2 (Moderate)= 50% ≤ FEV1 < 80% predicted; GOLD 3 (Severe) = 30% ≤ FEV1 < 50% predicted; GOLD 4 (Very Severe) = FEV1 < 30% predicted.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 4
Measure: Count of Units; unit: Sputum samples
Units Other Than Participants: Sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 197
Number analyzed (Sputum samples) | 280
Sputum samples
  Any, GOLD 2: number analyzed (Sputum samples) | 224
  Any, GOLD 2 | 150
  Any, GOLD 3 | 217
  Any, GOLD 4: number analyzed (Sputum samples) | 50
  Any, GOLD 4 | 44
  Hi, GOLD 2: number analyzed (Sputum samples) | 13
  Hi, GOLD 2 | 12
  Hi, GOLD 3: number analyzed (Sputum samples) | 21
  Hi, GOLD 3 | 20
  Hi, GOLD 4: number analyzed (Sputum samples) | 3
  Hi, GOLD 4 | 3
  NTHi, GOLD 2: number analyzed (Sputum samples) | 13
  NTHi, GOLD 2 | 12
  NTHi, GOLD 3: number analyzed (Sputum samples) | 21
  NTHi, GOLD 3 | 20
  NTHi, GOLD 4: number analyzed (Sputum samples) | 3
  NTHi, GOLD 4 | 3
  Non-Hi, GOLD 2: number analyzed (Sputum samples) | 13
  Non-Hi, GOLD 2 | 1
  Non-Hi, GOLD 3: number analyzed (Sputum samples) | 21
  Non-Hi, GOLD 3 | 1
  Non-Hi, GOLD 4: number analyzed (Sputum samples) | 3
  Non-Hi, GOLD 4 | 0
  M. catarrhalis, GOLD 2: number analyzed (Sputum samples) | 224
  M. catarrhalis, GOLD 2 | 0
  M. catarrhalis, GOLD 3 | 5
  M. catarrhalis, GOLD 4: number analyzed (Sputum samples) | 50
  M. catarrhalis, GOLD 4 | 0
  S. pneumoniae, GOLD 2: number analyzed (Sputum samples) | 224
  S. pneumoniae, GOLD 2 | 4
  S. pneumoniae, GOLD 3 | 10
  S. pneumoniae, GOLD 4: number analyzed (Sputum samples) | 50
  S. pneumoniae, GOLD 4 | 0
  S. aureus, GOLD 2: number analyzed (Sputum samples) | 224
  S. aureus, GOLD 2 | 7
  S. aureus, GOLD 3 | 6
  S. aureus, GOLD 4: number analyzed (Sputum samples) | 50
  S. aureus, GOLD 4 | 4
  P. aeruginosa, GOLD 2: number analyzed (Sputum samples) | 224
  P. aeruginosa, GOLD 2 | 14
  P. aeruginosa, GOLD 3 | 24
  P. aeruginosa, GOLD 4: number analyzed (Sputum samples) | 50
  P. aeruginosa, GOLD 4 | 9
  K. pneumoniae, GOLD 2: number analyzed (Sputum samples) | 224
  K. pneumoniae, GOLD 2 | 70
  K. pneumoniae, GOLD 3 | 60
  K. pneumoniae, GOLD 4: number analyzed (Sputum samples) | 50
  K. pneumoniae, GOLD 4 | 16
  A. baumannii, GOLD 2: number analyzed (Sputum samples) | 224
  A. baumannii, GOLD 2 | 2
  A. baumannii, GOLD 3: number analyzed (Sputum samples) | 279
  A. baumannii, GOLD 3 | 9
  A. baumannii, GOLD 4: number analyzed (Sputum samples) | 50
  A. baumannii, GOLD 4 | 1
  Other bacteria, GOLD 2: number analyzed (Sputum samples) | 224
  Other bacteria, GOLD 2 | 87
  Other bacteria, GOLD 3 | 149
  Other bacteria, GOLD 4: number analyzed (Sputum samples) | 50
  Other bacteria, GOLD 4 | 28

6. Secondary Outcome: Number of Sputum Samples Positive for Bacterial Pathogens (Overall and by Species) in Stable COPD Patients, as Identified by PCR, and Classified by GOLD Grade
Description: Number of sputum samples obtained at each confirmed stable visit, and positive for bacterial pathogens by PCR (overall and by bacterial species). The spirometric classification of airflow limitation in COPD patients is based on post-bronchodilator forced expiratory volume in 1 second (FEV1) and can be divided into four GOLD grades [GOLD, 2013]: GOLD 1 (MILD): FEV1 ≥ 80% predicted; GOLD 2 (Moderate)= 50% ≤ FEV1 < 80% predicted; GOLD 3 (Severe) = 30% ≤ FEV1 < 50% predicted; GOLD 4 (Very Severe) = FEV1 < 30% predicted.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 4
Measure: Count of Units; unit: Sputum samples
Units Other Than Participants: Sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 197
Number analyzed (Sputum samples) | 277
Sputum samples
  Any, GOLD 2: number analyzed (Sputum samples) | 221
  Any, GOLD 2 | 146
  Any, GOLD 3 | 184
  Any, GOLD 4: number analyzed (Sputum samples) | 48
  Any, GOLD 4 | 36
  H. influenzae, GOLD 2: number analyzed (Sputum samples) | 221
  H. influenzae, GOLD 2 | 95
  H. influenzae, GOLD 3 | 120
  H. influenzae, GOLD 4: number analyzed (Sputum samples) | 48
  H. influenzae, GOLD 4 | 19
  M. catarrhalis, GOLD 2: number analyzed (Sputum samples) | 221
  M. catarrhalis, GOLD 2 | 30
  M. catarrhalis, GOLD 3 | 42
  M. catarrhalis, GOLD 4: number analyzed (Sputum samples) | 48
  M. catarrhalis, GOLD 4 | 3
  S. pneumoniae, GOLD 2: number analyzed (Sputum samples) | 221
  S. pneumoniae, GOLD 2 | 39
  S. pneumoniae, GOLD 3 | 47
  S. pneumoniae, GOLD 4: number analyzed (Sputum samples) | 48
  S. pneumoniae, GOLD 4 | 6
  S. aureus, GOLD 2: number analyzed (Sputum samples) | 221
  S. aureus, GOLD 2 | 33
  S. aureus, GOLD 3 | 20
  S. aureus, GOLD 4: number analyzed (Sputum samples) | 48
  S. aureus, GOLD 4 | 5
  P. aeruginosa, GOLD 2: number analyzed (Sputum samples) | 221
  P. aeruginosa, GOLD 2 | 33
  P. aeruginosa, GOLD 3 | 44
  P. aeruginosa, GOLD 4: number analyzed (Sputum samples) | 48
  P. aeruginosa, GOLD 4 | 12
  S. pyogenes, GOLD 2: number analyzed (Sputum samples) | 221
  S. pyogenes, GOLD 2 | 1
  S. pyogenes, GOLD 3 | 1
  S. pyogenes, GOLD 4: number analyzed (Sputum samples) | 48
  S. pyogenes, GOLD 4 | 0

7. Secondary Outcome: Number of Sputum Samples Positive for Viral Pathogens (Overall and by Species) in Stable COPD Patients, as Identified by PCR, and Classified by GOLD Grade
Description: Number of sputum samples obtained at each confirmed stable visit, and positive for virus pathogens by PCR (overall and by viral species). The spirometric classification of airflow limitation in COPD patients is based on post-bronchodilator forced expiratory volume in 1 second (FEV1) and can be divided into four GOLD grades [GOLD, 2013]: GOLD 1 (MILD): FEV1 ≥ 80% predicted; GOLD 2 (Moderate)= 50% ≤ FEV1 < 80% predicted; GOLD 3 (Severe) = 30% ≤ FEV1 < 50% predicted; GOLD 4 (Very Severe) = FEV1 < 30% predicted.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 4
Measure: Count of Units; unit: Sputum samples
Units Other Than Participants: Sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 197
Number analyzed (Sputum samples) | 277
Sputum samples
  Any, GOLD 2: number analyzed (Sputum samples) | 221
  Any, GOLD 2 | 25
  Any, GOLD 3 | 52
  Any, GOLD 4: number analyzed (Sputum samples) | 48
  Any, GOLD 4 | 5
  RSV, GOLD 2: number analyzed (Sputum samples) | 221
  RSV, GOLD 2 | 1
  RSV, GOLD 3 | 3
  RSV, GOLD 4: number analyzed (Sputum samples) | 48
  RSV, GOLD 4 | 1
  Parainfluenza virus, GOLD 2: number analyzed (Sputum samples) | 221
  Parainfluenza virus, GOLD 2 | 1
  Parainfluenza virus, GOLD 3: number analyzed (Sputum samples) | 276
  Parainfluenza virus, GOLD 3 | 3
  Parainfluenza virus, GOLD 4: number analyzed (Sputum samples) | 48
  Parainfluenza virus, GOLD 4 | 0
  Enterovirus, GOLD 2: number analyzed (Sputum samples) | 221
  Enterovirus, GOLD 2 | 0
  Enterovirus, GOLD 3: number analyzed (Sputum samples) | 276
  Enterovirus, GOLD 3 | 3
  Enterovirus, GOLD 4: number analyzed (Sputum samples) | 48
  Enterovirus, GOLD 4 | 0
  HRV, GOLD 2: number analyzed (Sputum samples) | 221
  HRV, GOLD 2 | 14
  HRV, GOLD 3 | 27
  HRV, GOLD 4: number analyzed (Sputum samples) | 48
  HRV, GOLD 4 | 3
  Metapneumovirus, GOLD 2: number analyzed (Sputum samples) | 221
  Metapneumovirus, GOLD 2 | 0
  Metapneumovirus, GOLD 3: number analyzed (Sputum samples) | 276
  Metapneumovirus, GOLD 3 | 0
  Metapneumovirus, GOLD 4: number analyzed (Sputum samples) | 48
  Metapneumovirus, GOLD 4 | 0
  Influenza virus, GOLD 2: number analyzed (Sputum samples) | 221
  Influenza virus, GOLD 2 | 1
  Influenza virus, GOLD 3 | 3
  Influenza virus, GOLD 4: number analyzed (Sputum samples) | 48
  Influenza virus, GOLD 4 | 0
  Adenovirus, GOLD 2: number analyzed (Sputum samples) | 221
  Adenovirus, GOLD 2 | 6
  Adenovirus, GOLD 3: number analyzed (Sputum samples) | 276
  Adenovirus, GOLD 3 | 5
  Adenovirus, GOLD 4: number analyzed (Sputum samples) | 48
  Adenovirus, GOLD 4 | 0
  Bocavirus, GOLD 2: number analyzed (Sputum samples) | 221
  Bocavirus, GOLD 2 | 0
  Bocavirus, GOLD 3 | 1
  Bocavirus, GOLD 4: number analyzed (Sputum samples) | 48
  Bocavirus, GOLD 4 | 0
  Coronavirus, GOLD 2: number analyzed (Sputum samples) | 221
  Coronavirus, GOLD 2 | 2
  Coronavirus, GOLD 3 | 11
  Coronavirus, GOLD 4: number analyzed (Sputum samples) | 48
  Coronavirus, GOLD 4 | 1

8. Secondary Outcome: Number of Sputum Samples Positive for Bacterial Pathogens (Overall and by Species) in AECOPD Patients, as Identified by Bacteriological Methods and Classified by Severity of AECOPD
Description: Number of sputum samples obtained at each AECOPD visit, and positive for bacterial pathogens by bacteriological methods (overall and by bacterial species). Classification of severity of AECOPD as follows: Mild = controlled with an increase in dosage of regular medications; Moderate = requires treatment with systemic corticosteroids and/or antibiotics; Severe = requires hospitalization.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 4
Measure: Count of Units; unit: Sputum samples
Units Other Than Participants: Sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 88
Number analyzed (Sputum samples) | 209
Sputum samples
  Any, Mild AECOPD: number analyzed (Sputum samples) | 15
  Any, Mild AECOPD | 9
  Any, Moderate AECOPD: number analyzed (Sputum samples) | 171
  Any, Moderate AECOPD | 138
  Any, Severe AECOPD: number analyzed (Sputum samples) | 23
  Any, Severe AECOPD | 16
  Hi, Mild AECOPD: number analyzed (Sputum samples) | 3
  Hi, Mild AECOPD | 3
  Hi, Moderate AECOPD: number analyzed (Sputum samples) | 12
  Hi, Moderate AECOPD | 11
  Hi, Severe AECOPD: number analyzed (Sputum samples) | 2
  Hi, Severe AECOPD | 2
  NTHi, Mild AECOPD: number analyzed (Sputum samples) | 3
  NTHi, Mild AECOPD | 3
  NTHi, Moderate AECOPD: number analyzed (Sputum samples) | 12
  NTHi, Moderate AECOPD | 11
  NTHi, Severe AECOPD: number analyzed (Sputum samples) | 2
  NTHi, Severe AECOPD | 2
  Non-Hi, Mild AECOPD: number analyzed (Sputum samples) | 3
  Non-Hi, Mild AECOPD | 0
  Non-Hi, Moderate AECOPD: number analyzed (Sputum samples) | 12
  Non-Hi, Moderate AECOPD | 1
  Non-Hi, Severe AECOPD: number analyzed (Sputum samples) | 2
  Non-Hi, Severe AECOPD | 0
  M. catarrhalis, Mild AECOPD: number analyzed (Sputum samples) | 15
  M. catarrhalis, Mild AECOPD | 0
  M. catarrhalis, Moderate AECOPD: number analyzed (Sputum samples) | 171
  M. catarrhalis, Moderate AECOPD | 6
  M. catarrhalis, Severe AECOPD: number analyzed (Sputum samples) | 23
  M. catarrhalis, Severe AECOPD | 1
  S. pneumoniae, Mild AECOPD: number analyzed (Sputum samples) | 15
  S. pneumoniae, Mild AECOPD | 0
  S. pneumoniae, Moderate AECOPD: number analyzed (Sputum samples) | 171
  S. pneumoniae, Moderate AECOPD | 5
  S. pneumoniae, Severe AECOPD: number analyzed (Sputum samples) | 23
  S. pneumoniae, Severe AECOPD | 0
  S. aureus, Mild AECOPD: number analyzed (Sputum samples) | 15
  S. aureus, Mild AECOPD | 0
  S. aureus, Moderate AECOPD: number analyzed (Sputum samples) | 171
  S. aureus, Moderate AECOPD | 5
  S. aureus, Severe AECOPD: number analyzed (Sputum samples) | 23
  S. aureus, Severe AECOPD | 2
  P. aeruginosa, Mild AECOPD: number analyzed (Sputum samples) | 15
  P. aeruginosa, Mild AECOPD | 1
  P. aeruginosa, Moderate AECOPD: number analyzed (Sputum samples) | 171
  P. aeruginosa, Moderate AECOPD | 26
  P. aeruginosa, Severe AECOPD: number analyzed (Sputum samples) | 23
  P. aeruginosa, Severe AECOPD | 3
  K. pneumoniae, Mild AECOPD: number analyzed (Sputum samples) | 15
  K. pneumoniae, Mild AECOPD | 4
  K. pneumoniae, Moderate AECOPD: number analyzed (Sputum samples) | 171
  K. pneumoniae, Moderate AECOPD | 43
  K. pneumoniae, Severe AECOPD: number analyzed (Sputum samples) | 23
  K. pneumoniae, Severe AECOPD | 5
  A. baumannii, Mild AECOPD: number analyzed (Sputum samples) | 15
  A. baumannii, Mild AECOPD | 1
  A. baumannii, Moderate AECOPD: number analyzed (Sputum samples) | 171
  A. baumannii, Moderate AECOPD | 8
  A. baumannii, Severe AECOPD: number analyzed (Sputum samples) | 23
  A. baumannii, Severe AECOPD | 0
  Other bacteria, Mild AECOPD: number analyzed (Sputum samples) | 15
  Other bacteria, Mild AECOPD | 4
  Other bacteria, Moderate AECOPD: number analyzed (Sputum samples) | 171
  Other bacteria, Moderate AECOPD | 84
  Other bacteria, Severe AECOPD: number analyzed (Sputum samples) | 23
  Other bacteria, Severe AECOPD | 6

9. Secondary Outcome: Number of Sputum Samples Positive for Bacterial Pathogens (Overall and by Species) in AECOPD Patients, as Identified by PCR, and Classified by Severity of AECOPD
Description: Number of sputum samples obtained at each AECOPD visit, and positive for bacterial pathogens by PCR (overall and by bacterial species). Classification of severity of AECOPD is as follows: Mild = controlled with an increase in dosage of regular medications; Moderate = requires treatment with systemic corticosteroids and/or antibiotics; Severe = requires hospitalization.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 4
Measure: Count of Units; unit: Sputum samples
Units Other Than Participants: Sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 88
Number analyzed (Sputum samples) | 194
Sputum samples
  Any, Mild AECOPD: number analyzed (Sputum samples) | 15
  Any, Mild AECOPD | 13
  Any, Moderate AECOPD: number analyzed (Sputum samples) | 157
  Any, Moderate AECOPD | 117
  Any, Severe AECOPD: number analyzed (Sputum samples) | 22
  Any, Severe AECOPD | 15
  H. influenzae, Mild AECOPD: number analyzed (Sputum samples) | 15
  H. influenzae, Mild AECOPD | 10
  H. influenzae, Moderate AECOPD: number analyzed (Sputum samples) | 157
  H. influenzae, Moderate AECOPD | 62
  H. influenzae, Severe AECOPD: number analyzed (Sputum samples) | 22
  H. influenzae, Severe AECOPD | 5
  M. catarrhalis, Mild AECOPD: number analyzed (Sputum samples) | 15
  M. catarrhalis, Mild AECOPD | 3
  M. catarrhalis, Moderate AECOPD: number analyzed (Sputum samples) | 157
  M. catarrhalis, Moderate AECOPD | 44
  M. catarrhalis, Severe AECOPD: number analyzed (Sputum samples) | 22
  M. catarrhalis, Severe AECOPD | 5
  S. pneumoniae, Mild AECOPD: number analyzed (Sputum samples) | 15
  S. pneumoniae, Mild AECOPD | 1
  S. pneumoniae, Moderate AECOPD: number analyzed (Sputum samples) | 157
  S. pneumoniae, Moderate AECOPD | 32
  S. pneumoniae, Severe AECOPD: number analyzed (Sputum samples) | 22
  S. pneumoniae, Severe AECOPD | 4
  S. aureus, Mild AECOPD: number analyzed (Sputum samples) | 15
  S. aureus, Mild AECOPD | 1
  S. aureus, Moderate AECOPD: number analyzed (Sputum samples) | 157
  S. aureus, Moderate AECOPD | 15
  S. aureus, Severe AECOPD: number analyzed (Sputum samples) | 22
  S. aureus, Severe AECOPD | 2
  P. aeruginosa, Mild AECOPD: number analyzed (Sputum samples) | 15
  P. aeruginosa, Mild AECOPD | 2
  P. aeruginosa, Moderate AECOPD: number analyzed (Sputum samples) | 157
  P. aeruginosa, Moderate AECOPD | 24
  P. aeruginosa, Severe AECOPD: number analyzed (Sputum samples) | 22
  P. aeruginosa, Severe AECOPD | 6
  S. pyogenes, Mild AECOPD: number analyzed (Sputum samples) | 15
  S. pyogenes, Mild AECOPD | 0
  S. pyogenes, Moderate AECOPD: number analyzed (Sputum samples) | 157
  S. pyogenes, Moderate AECOPD | 2
  S. pyogenes, Severe AECOPD: number analyzed (Sputum samples) | 22
  S. pyogenes, Severe AECOPD | 0

10. Secondary Outcome: Number of Sputum Samples Positive for Viral Pathogens (Overall and by Species) in AECOPD Patients, as Identified by PCR, and Classified by Severity of AECOPD
Description: Number of sputum samples obtained at each AECOPD visit, and positive for viral pathogens by PCR (overall and by viral species). Classification of severity of AECOPD is as follows: Mild = controlled with an increase in dosage of regular medications; Moderate = requires treatment with systemic corticosteroids and/or antibiotics; Severe = requires hospitalization.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 4
Measure: Count of Units; unit: Sputum samples
Units Other Than Participants: Sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 88
Number analyzed (Sputum samples) | 194
Sputum samples
  Any, Mild AECOPD: number analyzed (Sputum samples) | 15
  Any, Mild AECOPD | 6
  Any, Moderate AECOPD: number analyzed (Sputum samples) | 157
  Any, Moderate AECOPD | 56
  Any, Severe AECOPD: number analyzed (Sputum samples) | 22
  Any, Severe AECOPD | 7
  RSV, Mild AECOPD: number analyzed (Sputum samples) | 15
  RSV, Mild AECOPD | 1
  RSV, Moderate AECOPD: number analyzed (Sputum samples) | 157
  RSV, Moderate AECOPD | 1
  RSV, Severe AECOPD: number analyzed (Sputum samples) | 22
  RSV, Severe AECOPD | 0
  Parainfluenza virus, Mild AECOPD: number analyzed (Sputum samples) | 15
  Parainfluenza virus, Mild AECOPD | 1
  Parainfluenza virus, Moderate AECOPD: number analyzed (Sputum samples) | 156
  Parainfluenza virus, Moderate AECOPD | 6
  Parainfluenza virus, Severe AECOPD: number analyzed (Sputum samples) | 22
  Parainfluenza virus, Severe AECOPD | 2
  Enterovirus, Mild AECOPD: number analyzed (Sputum samples) | 15
  Enterovirus, Mild AECOPD | 0
  Enterovirus, Moderate AECOPD: number analyzed (Sputum samples) | 156
  Enterovirus, Moderate AECOPD | 0
  Enterovirus, Severe AECOPD: number analyzed (Sputum samples) | 22
  Enterovirus, Severe AECOPD | 0
  HRV, Mild AECOPD: number analyzed (Sputum samples) | 15
  HRV, Mild AECOPD | 3
  HRV, Moderate AECOPD: number analyzed (Sputum samples) | 157
  HRV, Moderate AECOPD | 26
  HRV, Severe AECOPD: number analyzed (Sputum samples) | 22
  HRV, Severe AECOPD | 3
  Metapneumovirus, Mild AECOPD: number analyzed (Sputum samples) | 15
  Metapneumovirus, Mild AECOPD | 0
  Metapneumovirus, Moderate AECOPD: number analyzed (Sputum samples) | 156
  Metapneumovirus, Moderate AECOPD | 0
  Metapneumovirus, Severe AECOPD: number analyzed (Sputum samples) | 22
  Metapneumovirus, Severe AECOPD | 0
  Influenza virus, Mild AECOPD: number analyzed (Sputum samples) | 15
  Influenza virus, Mild AECOPD | 1
  Influenza virus, Moderate AECOPD: number analyzed (Sputum samples) | 157
  Influenza virus, Moderate AECOPD | 14
  Influenza virus, Severe AECOPD: number analyzed (Sputum samples) | 22
  Influenza virus, Severe AECOPD | 1
  Adenovirus, Mild AECOPD: number analyzed (Sputum samples) | 15
  Adenovirus, Mild AECOPD | 0
  Adenovirus, Moderate AECOPD: number analyzed (Sputum samples) | 156
  Adenovirus, Moderate AECOPD | 7
  Adenovirus, Severe AECOPD: number analyzed (Sputum samples) | 22
  Adenovirus, Severe AECOPD | 1
  Bocavirus, Mild AECOPD: number analyzed (Sputum samples) | 15
  Bocavirus, Mild AECOPD | 0
  Bocavirus, Moderate AECOPD: number analyzed (Sputum samples) | 157
  Bocavirus, Moderate AECOPD | 0
  Bocavirus, Severe AECOPD: number analyzed (Sputum samples) | 22
  Bocavirus, Severe AECOPD | 0
  Coronavirus, Mild AECOPD: number analyzed (Sputum samples) | 15
  Coronavirus, Mild AECOPD | 1
  Coronavirus, Moderate AECOPD: number analyzed (Sputum samples) | 157
  Coronavirus, Moderate AECOPD | 9
  Coronavirus, Severe AECOPD: number analyzed (Sputum samples) | 22
  Coronavirus, Severe AECOPD | 1

11. Secondary Outcome: Incidence Rate (Per Subject Per Year) of Confirmed and Confirmed Plus Potential AECOPDs, Overall and by GOLD Grade
Description: Incidence rate is estimated by the mean number of exacerbations per subject and per year from Negative Binomial model (or Poisson model in case of under dispersion) without covariates and computed with 95% confidence intervals (CI). Confirmed AECOPDs include AECOPD events plus missed AECOPD events (i.e.: all morning alerts confirmed by phone call (as well as cases with no morning alert) for which there has been no site visit but for which AECOPD medical records are available). Potential AECOPDs include all morning alert confirmed by phone call for which there has been no site visit and for which no medical records are available.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: AECOPDs per person-year
Arm/Group | Total Group
Number analyzed (Participants) | 197
AECOPDs per person-year
  Total, Confirmed AECOPDs | 1.27 [1.04 to 1.54]
  GOLD 2, Confirmed AECOPDs: number analyzed (Participants) | 79
  GOLD 2, Confirmed AECOPDs | 0.78 [0.54 to 1.14]
  GOLD 3, Confirmed AECOPDs: number analyzed (Participants) | 99
  GOLD 3, Confirmed AECOPDs | 1.51 [1.17 to 1.94]
  GOLD 4, Confirmed AECOPDs: number analyzed (Participants) | 19
  GOLD 4, Confirmed AECOPDs | 1.99 [1.37 to 2.89]
  Total, Confirmed AECOPDs plus potential AECOPDs | 1.3 [1.07 to 1.58]
  GOLD 2, Confirmed AECOPDs plus potential AECOPDs: number analyzed (Participants) | 79
  GOLD 2, Confirmed AECOPDs plus potential AECOPDs | 0.81 [0.56 to 1.16]
  GOLD 3, Confirmed AECOPDs plus potential AECOPDs: number analyzed (Participants) | 99
  GOLD 3, Confirmed AECOPDs plus potential AECOPDs | 1.56 [1.20 to 2.01]
  GOLD 4, Confirmed AECOPDs plus potential AECOPDs: number analyzed (Participants) | 19
  GOLD 4, Confirmed AECOPDs plus potential AECOPDs | 1.99 [1.37 to 2.89]

12. Secondary Outcome: Number of Subjects With AECOPDs, Classified by Number of Exacerbations and by Severity of AECOPD
Description: Classification of severity of AECOPD is as follows: Mild- Controlled AECOPD with an increase in dosage of regular medications; Moderate- Requires treatment with systemic corticosteroids and/ or antibiotics; Severe- Requires hospitalisation.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 197
Participants
  Mild AECOPD, 0 | 181
  Moderate AECOPD, 0 | 115
  Severe AECOPD, 0 | 168
  Mild AECOPD, 1 | 12
  Moderate AECOPD, 1 | 38
  Severe AECOPD, 1 | 21
  Mild AECOPD, 2 | 3
  Moderate AECOPD, 2 | 15
  Severe AECOPD, 2 | 7
  Mild AECOPD, 3 | 1
  Moderate AECOPD, 3 | 11
  Severe AECOPD, 3 | 0
  Mild AECOPD, 4 | 0
  Moderate AECOPD, 4 | 7
  Severe AECOPD, 4 | 1
  Mild AECOPD, >4 | 0
  Moderate AECOPD, >4 | 11
  Severe AECOPD, >4 | 0

13. Secondary Outcome: Number of Subjects With AECOPDs, Classified by Number of Exacerbations and by GOLD Grade
Description: The spirometric classification of airflow limitation in COPD patients is based on post-bronchodilator forced expiratory volume in 1 second (FEV1) and can be divided into four GOLD grades [GOLD, 2013]: GOLD 1 (MILD): FEV1 ≥ 80% predicted; GOLD 2 (Moderate)= 50% ≤ FEV1 < 80% predicted; GOLD 3 (Severe) = 30% ≤ FEV1 < 50% predicted; GOLD 4 (Very Severe) = FEV1 < 30% predicted.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 99
Participants
  GOLD 2, 0: number analyzed (Participants) | 79
  GOLD 2, 0 | 48
  GOLD 2, 1: number analyzed (Participants) | 79
  GOLD 2, 1 | 17
  GOLD 2, 2: number analyzed (Participants) | 79
  GOLD 2, 2 | 6
  GOLD 2, 3: number analyzed (Participants) | 79
  GOLD 2, 3 | 4
  GOLD 2, 4: number analyzed (Participants) | 79
  GOLD 2, 4 | 1
  GOLD 2, >4: number analyzed (Participants) | 79
  GOLD 2, >4 | 3
  GOLD 3, 0 | 42
  GOLD 3, 1 | 15
  GOLD 3, 2 | 21
  GOLD 3, 3 | 5
  GOLD 3, 4 | 7
  GOLD 3, >4 | 9
  GOLD 4, 0: number analyzed (Participants) | 19
  GOLD 4, 0 | 3
  GOLD 4, 1: number analyzed (Participants) | 19
  GOLD 4, 1 | 6
  GOLD 4, 2: number analyzed (Participants) | 19
  GOLD 4, 2 | 5
  GOLD 4, 3: number analyzed (Participants) | 19
  GOLD 4, 3 | 0
  GOLD 4, 4: number analyzed (Participants) | 19
  GOLD 4, 4 | 4
  GOLD 4, >4: number analyzed (Participants) | 19
  GOLD 4, >4 | 1

14. Secondary Outcome: Number of Days of AECOPD Episodes, Overall and by AECOPD Severity
Description: Descriptive statistics (mean, standard deviation) on the number of days of AECOPD episodes are presented, overall and by AECOPD severity.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Total Group
Number analyzed (Participants) | 227
Days
  Any Severity | 14.3 (9.0)
  Mild: number analyzed (Participants) | 21
  Mild | 20.3 (11.1)
  Moderate: number analyzed (Participants) | 182
  Moderate | 12.6 (6.3)
  Severe: number analyzed (Participants) | 24
  Severe | 21.5 (16.5)

15. Secondary Outcome: COPD Assessment Test (CAT) Score in Stable COPD Patients
Description: The CAT is a patient-completed instrument to assess the heath-related quality of life (HRQOL) and symptom burden in patients with COPD. Descriptive statistics (mean, standard deviation) on the CAT scores are tabulated at each stable visit. The CAT index is derived as the sum of the ratings recorded for each of the eight individual items. Each of these items has 6 possible scores (0, 1, 2, 3, 4 or 5), leading to a range of 0 (best score) to 40 (worst score) for CAT score.
Time Frame: At Month 0, Month 6 and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on the CAT scale
Arm/Group | Total Group
Number analyzed (Participants) | 197
Units on the CAT scale
  Month 0 | 11.78 (5.56)
  Month 6: number analyzed (Participants) | 186
  Month 6 | 12.56 (6.08)
  Month 12: number analyzed (Participants) | 181
  Month 12 | 13.71 (6.53)

16. Secondary Outcome: CAT Score by Frequency of Exacerbations
Description: The CAT is a patient-completed instrument to assess the HRQOL and symptom burden in patients with COPD. Descriptive statistics (mean, standard deviation) on the CAT scores are tabulated by frequency of exacerbations). The CAT index is derived as the sum of the ratings recorded for each of the eight individual items. Each of these items has 6 possible scores (0, 1, 2, 3, 4 or 5), leading to a range of 0 (best score) to 40 (worst score) for CAT score.
Time Frame: Over the course of one year from the study start: (Month 0 to Month 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on the CAT scale
Arm/Group | Total Group
Number analyzed (Participants) | 41
Units on the CAT scale
  1 exacerbation: number analyzed (Participants) | 38
  1 exacerbation | 2.05 (5.62)
  2 or 3 exacerbations | 3.08 (5.01)
  >3 exacerbations: number analyzed (Participants) | 25
  >3 exacerbations | 3.79 (4.84)

17. Secondary Outcome: St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) Score in Stable COPD Patients
Description: The SGRQ-C is designed to assess HRQOL and current health of the patients. Descriptive statistics (mean, standard deviation) on the SGRQ-C scores are tabulated at each stable visit. The SGRQ-C total score is derived as the weighted sum of the forty individual items leading to a range of 0 (best score) to 100 (worst score) as detailed in the reference manual [St George's Respiratory Questionnaire for COPD patients, version 1.3, 2016].
Time Frame: At Month 0, Month 6 and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on the SGRQ-C scale
Arm/Group | Total Group
Number analyzed (Participants) | 197
Units on the SGRQ-C scale
  Month 0 | 35.22 (17.21)
  Month 6: number analyzed (Participants) | 184
  Month 6 | 34.38 (16.52)
  Month 12: number analyzed (Participants) | 178
  Month 12 | 35.1 (17.86)

18. Secondary Outcome: Post-bronchodilator FEV1 Percentage of Predicted Normal Value in Stable COPD Patients
Description: Summary statistics (mean, standard deviation) on post bronchodilator FEV1% of predicted normal value is tabulated at enrolment and final visit.
Time Frame: At Pre-Month 0 (screening visit) and Month 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of FEV1
Arm/Group | Total Group
Number analyzed (Participants) | 197
Percentage of FEV1
  Pre-Month 0 | 47.83 (13.94)
  Month 12 | 46.93 (14.93)

19. Secondary Outcome: Number of Patients With Healthcare Utilisation During Stable Periods
Description: Healthcare utilization includes all unscheduled visits to a physician office, visits to urgent care, visits to emergency department, and hospitalizations. The impact of AECOPD on healthcare utilization is assessed during the stable periods. Hospitalizations that were associated with the disease being studied were not collected as Adverse Events (AEs) or as serious AEs (SAEs) as per protocol.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 197
Participants
  Physician's office consultations | 135
  Urgent care | 4
  Emergency department | 20
  Hospitalization | 26

20. Secondary Outcome: Number of Patients With Healthcare Utilisation During Exacerbation Periods
Description: Healthcare utilization includes all unscheduled visits to a physician office, visits to urgent care, visits to emergency department, and hospitalizations. The impact of AECOPD on healthcare utilization is assessed during exacerbation periods. Hospitalizations that were associated with the disease being studied were not collected as AEs or as SAEs as per protocol.
Time Frame: Over the course of one year from the study start (Month 0 to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 104
Participants
  Physician's office consultations | 48
  Urgent care | 2
  Emergency department | 13
  Hospitalization | 20

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events and serious adverse events (SAE) related to study procedures have been collected during the whole study period (from Month 0 to Month 12.
Description: In the Participant flow section, there are 2 participants reported with "adverse event" reason for not completed: 1 was for SAE described in the Serious Adverse Events section below, and the other one was for a SAE not related to study procedure, and hence, no information (System Organ Class & Preferred Term) was collected, as per protocol, for this SAE. Hospitalizations that were associated with the disease being studied were not collected as AEs or as SAEs as per protocol.
Arm/Group | Total Group
All-Cause Mortality (participants affected / at risk) | 2/197
Serious Adverse Events (participants affected / at risk) | 1/197
Other Adverse Events (participants affected / at risk) | 1/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Group (N=197)
Pneumonia necrotizing (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Group (N=197)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT03151395/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT03151395/SAP_001.pdf